CLINICAL TRIAL: NCT05919303
Title: Multidetector Computed Tomography (MDCT) Evaluation of Obstructive Jaundice: A Cross-sectional Study From a Tertiary Hospital of Nepal
Status: Completed | Type: Observational
Sponsor: Shree Birendra Hospital (Other)
Collaborators: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Asim Mahat, Doctor, Shree Birendra Hospital
Other Study IDs: Acd/291/075/076-IRC
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Obstuctive Jaundice; Radiological Correlation of Obstructive Jaundice

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient presenting with obstructive jaundice referred for CT evaluation
  Interventions: Radiation: CT Scan

INTERVENTIONS:
Radiation: CT Scan — CT scan study of abdomen

SUMMARY:
This study was done to evaluate the diagnostic statistics of MDCT and its features in the assessment of obstructive jaundice in reference to surgical or histopathological diagnosis.

DETAILED DESCRIPTION:
We did a cross-sectional study among 30 participants of obstructive jaundice at BP Koirala Institute of Health Sciences (BPKIHS), Dharan, Nepal. The sensitivity and the Negative predictive value of MDCT for non-neoplastic cause to detect obstructive jaundice were 100% (95% CI 79.41-100.00) and 100% (95% CI 75.29-100.00), while the specificity and the Positive predictive value for neoplastic cause to detect obstructive jaundice were 100% (95% CI: 79.41-100.00) and 100% (95% CI: 75.29-100.00). Similarly, the accuracy for either non-neoplastic or neoplastic cause was 96.67% (95% CI: 82.78-99.92). The most common cause for obstructive jaundice was choledocholithiasis (33.34%) followed by cholangiocarcinoma (20%), ampullary carcinoma (13.33%) and choledochal cyst (13.33%). The diagnostic accuracy of individual etiology of common causes of obstructive jaundice ranged from 82.78 to 100%. Biliary obstruction was most frequently observed in the periampullary region (83.33%), followed by the proximal common bile duct (6.67%), hilar region (6.67%), and intrahepatic region (3.33%).The MDCT could serve as the initial, cost-effective, easily available, and time-efficient imaging modality for diagnosing various causes of obstructive jaundice. It can differentiate non-neoplastic from neoplastic causes of obstructive jaundice.

ELIGIBILITY:
Inclusion Criteria:

* Any patient referred for CT scan with findings suggestive of obstructive jaundice with pertinent Histopathological and post-surgical findings .

Exclusion Criteria:

* Patients with contraindications for contrast-enhanced CT, those with non-obstructive cases of jaundice, and patients experiencing recurrent malignancy causing obstructive jaundice.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 30 All patients exhibiting clinical and biochemical features of obstructive jaundice who were referred for MDCT scan and subsequently received a final diagnosis through histopathology, cytopathology or surgical findings were included as participants in the study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the diagnostic statistics of MDCT and its features in the assessment of obstructive jaundice in reference to surgical or histopathological diagnosis. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Asim Mahat, MD, Principal Investigator — Nepalese Army Institute of Health Sciences
Locations (1):
- BP Koirala Institute of Health Sciences, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: No